CLINICAL TRIAL: NCT04599075
Title: Intravenous Insulin Versus Subcutaneous Insulin Infusion in Intrapartum Management of Pregnant Women With Type 1 Diabetes Mellitus: A Randomized Trial
Brief Title: Intravenous Insulin vs Subcutaneous Insulin Infusion in Intrapartum Management of Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gianna Wilkie (Other)
Responsible Party: Sponsor-Investigator, Gianna Wilkie, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00021746
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes; Pregnancy, High Risk
Keywords: Pregnancy; Type 1 Diabetes; Intrapartum Insulin; Maternal Outcomes; Neonatal Outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized study evaluating intrapartum insulin delivery management strategies among pregnant women with type 1 diabetes mellitus.
Who Masked: Outcomes Assessor
Masking Description: Those assessing the outcomes from the medical chart will be blinded to the randomization process and the assigned study arm. Patients, the primary investigator, and their care providers will be aware of their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous Insulin Infusion (Experimental): Patients will be randomized to discontinuation of the CSII pump intrapartum and initiation of IV insulin infusion per hospital protocol.
  Interventions: Drug: Insulin
- Continuous Subcutaneous Insulin Infusion (CSII) (Experimental): Patients will be randomized to continuation of their CSII pump intrapartum and will be managed in accordance with the CSII hospital protocol.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — IV Insulin Infusion
  Other Names: Insulin via IV Infusion
  Arms: Intravenous Insulin Infusion
Drug: Insulin — Continuous Subcutaneous Insulin Infusion (Pump)
  Other Names: Insulin via Pump
  Arms: Continuous Subcutaneous Insulin Infusion (CSII)

SUMMARY:
The purpose of this study is to perform a randomized trial to investigate if intrapartum insulin delivery mechanisms reduces adverse outcomes associated with type 1 diabetes in pregnancy. The investigators aim to compare subcutaneous insulin pump versus intravenous insulin infusion with regard to the primary outcome of neonatal blood sugar.

DETAILED DESCRIPTION:
Intrapartum glucose management is critical to reducing neonatal hypoglycemia shortly after birth. Some providers are comfortable continuing patients on their subcutaneous insulin pump during labor while others transition these patients to intravenous insulin infusions. Previous literature has retrospectively shown this to be both a feasible and safe option.

The investigators aim to compare subcutaneous insulin pump versus intravenous insulin infusion with regard to obstetric and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with pre-gestational diagnosis of type 1 diabetes mellitus and managed on an insulin pump in pregnancy
* Pregnancy and delivery care obtained at University of Massachusetts (UMass) Memorial Medical Center
* Patients able to provide written informed consent

Exclusion Criteria:

* Patients who are under the age of 18
* Patients with altered state of consciousness
* Critically ill patient requiring intensive care unit admission
* Patient at risk for suicide
* Patient refuses or is otherwise unable to participate in own care
* Patient without pump supplies
* Patients presenting with diabetic ketoacidosis on admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianna L Wilkie, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldberg D, Dicker D, Samuel N, Peleg D, Karp M, Goldman JA. Intrapartum management of insulin-dependent diabetes mellitus (IDDM) gestants. A comparative study of constant intravenous insulin infusion and continuous subcutaneous insulin infusion pump (CSIIP). Acta Obstet Gynecol Scand. 1988;67(4):333-8. PMID 3051881
- [Background] Peterson C, Grosse SD, Li R, Sharma AJ, Razzaghi H, Herman WH, Gilboa SM. Preventable health and cost burden of adverse birth outcomes associated with pregestational diabetes in the United States. Am J Obstet Gynecol. 2015 Jan;212(1):74.e1-9. doi: 10.1016/j.ajog.2014.09.009. Epub 2014 Oct 28. PMID 25439811
- [Background] Professional Practice Committee for the Standards of Medical Care in Diabetes-2016. Diabetes Care. 2016 Jan;39 Suppl 1:S107-8. doi: 10.2337/dc16-S018. No abstract available. PMID 26696673
- [Background] Drever E, Tomlinson G, Bai AD, Feig DS. Insulin pump use compared with intravenous insulin during labour and delivery: the INSPIRED observational cohort study. Diabet Med. 2016 Sep;33(9):1253-9. doi: 10.1111/dme.13106. Epub 2016 Mar 20. PMID 26927202
- [Background] Fresa R, Visalli N, Di Blasi V, Cavallaro V, Ansaldi E, Trifoglio O, Abbruzzese S, Bongiovanni M, Agrusta M, Napoli A. Experiences of continuous subcutaneous insulin infusion in pregnant women with type 1 diabetes during delivery from four Italian centers: a retrospective observational study. Diabetes Technol Ther. 2013 Apr;15(4):328-34. doi: 10.1089/dia.2012.0260. Epub 2013 Mar 28. PMID 23537417
- [Derived] Wilkie GL, Delpapa E, Leftwich HK. Intrapartum continuous subcutaneous insulin infusion vs intravenous insulin infusion among pregnant individuals with type 1 diabetes mellitus: a randomized controlled trial. Am J Obstet Gynecol. 2023 Dec;229(6):680.e1-680.e8. doi: 10.1016/j.ajog.2023.07.003. Epub 2023 Jul 8. PMID 37429432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The row summary is the mean age and standard deviation.
  years | 29.2 (5.4) | 31.6 (4.7) | 30.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Nulliparous [Count of Participants; unit: Participants] | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Hypoglycemia
Description: First neonatal blood sugar obtained within 2 hours of birth
Time Frame: Within 2 hours of birth
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
mg/dL | 49.2 (22.6) | 50.1 (23.4)

2. Secondary Outcome: Number of Maternal Hypoglycemic Events
Description: Number of maternal blood sugars < 60 mg/dL
Time Frame: During labor
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 5 | 1

3. Secondary Outcome: Development of Diabetic Ketoacidosis During Labor
Description: Development of Diabetic Ketoacidosis during labor
Time Frame: During Labor
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

4. Secondary Outcome: Mode of Delivery
Description: Mode of Delivery (vaginal versus cesarean)
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants
  Cesarean Delivery | 17 | 23
  Vaginal | 16 | 11
  Operative Vaginal | 2 | 1

5. Secondary Outcome: Neonatal Birthweight
Description: Neonatal Birthweight
Time Frame: At Birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
grams | 3067.8 (1035.8) | 3293.3 (883.7)

6. Secondary Outcome: Number of Participants With Shoulder Dystocia
Description: Number of participants with shoulder dystocia
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 4 | 1

7. Secondary Outcome: Number of Participants With Brachial Plexus Injury
Description: Number of participants with brachial plexus injury
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

8. Secondary Outcome: 5 Minute Apgar Score < 7
Description: Neonatal Apgar Score: The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: At delivery (5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 7 | 3

9. Secondary Outcome: Received Neonatal Intervention for Hypoglycemia
Description: Received intervention for hypoglycemia (any oral, IV, or both)
Time Frame: Within 24 hours of life
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 18 | 20

10. Secondary Outcome: Neonatal Intensive Care Unit Admission
Description: Admission to level 2 or greater neonatal ICU. This is a marker for additional need for neonatal support and care after delivery.
Time Frame: At delivery and within first 2 day of life
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 16 | 17

11. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery
Time Frame: At birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
weeks | 35.6 (3.6) | 36.0 (2.8)

12. Secondary Outcome: Number of Participants With Neonatal Respiratory Distress
Description: Requiring 2 or more hours of respiratory support or oxygen with associated diagnosis
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 4 | 2

13. Secondary Outcome: Number of Participants With Neonatal Hyperbilirubinemia
Description: Requiring phototherapy
Time Frame: Within first 2 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
Number analyzed (Participants) | 35 | 35
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Intrapartum (on admission to labor and delivery) and for 24 hours postpartum)
Arm/Group | Intravenous Insulin Infusion | Continuous Subcutaneous Insulin Infusion (CSII)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT04599075/Prot_SAP_000.pdf